CLINICAL TRIAL: NCT05408377
Title: Effectiveness of Acupuncture for Cyclical Mastalgia （CM）
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pinggu Hospital of Beijing Traditional Chinese Medicine Hospital (Other)
Collaborators: Pinggu huangsongyu Community hospital (Unknown); Pinggu Xiagezhuang Community hospital (Unknown)
Responsible Party: Principal Investigator, Chuan Yu, Principal Investigator, Pinggu Hospital of Beijing Traditional Chinese Medicine Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CFH2022-3-7132
Record Dates: First submitted 2022-05-23; First posted 2022-06-07 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Mastalgia
Keywords: mastalgia
MeSH Terms: conditions — Mastodynia

STUDY DESIGN:
Intervention Model Description: This study is a 2-arm randomized controlled trial. According to the ratio of 1：1 and block randomization, a total of 108 eligible CM patients will be randomly allocated to either MA(n=54) or SA(n=54).
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Considering the particularity of acupuncture manipulation, acupuncturists in this trial cannot be blinded. The patients, evaluators, and statistical analysts will be blinded to the group allocation. The manipulation of needles will be similar in both groups. Unblinding will only be performed in cases of an emergency event.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MA group (Experimental): Manual Acupuncture
  Interventions: Other: MA group
- SA group (Placebo Comparator): Sham acupuncture
  Interventions: Other: SA group

INTERVENTIONS:
Other: MA group — We will select Ashi points (the most obvious local pain over the breast), Tanzhong(CV17), bilateral Wuyi (ST15), Rugen (ST18), Tianzong(SI11), Geshu (BL17), Ganshu(BL18), Hegu(LI4), Sanyinjiao (SP6) and Taichong (LR3)in this trial.After insertion, all needles will be manually manipulated (equal manipulations of twirling, lifting, and thrusting)to achieve De qi sensation.
  Arms: MA group
Other: SA group — The SA group will use a special needle in which the tip is blunt and the pedestal is opaque. There is an adhesive pad below the base to ensure that the whole pedestal can adhere to the points. Participants will receive superficial touch at bilateral sham GV8(Jinsuo), sham GV7(Zhongshu), sham GV6(Jizhong), sham GV5(Xuanshu), sham GV4(Mingmen), sham BL37(Yinmen), and sham BL57(Chengshan), the needles will touch the skin and not be inserted into the skin, then lift and twist each point evenly for 3 times, make the subject feel the similar sensation of deqi.
  Arms: SA group

SUMMARY:
This study is a multi-center 2-arm randomized controlled trial. According to the ratio of 1：1 and block randomization, a total of 108 eligible CM patients will be randomly allocated to either MA(n=54) or SA(n=54). All patients will undergo treatment two weeks before menstruation and treatment will be stopped at the onset of menstruation. Three times a week, six times a menstrual cycle, 3consecutive menstrual cycles for a total of 18 sessions after baseline. The primary outcome will be the change in the average daily breast pain VAS(VAS-BP) scores during the first 2 weeks of menstruation from baseline at weeks 4,8,12. Additionally, VAS-BP scores at weeks 24 and 36 will also be assessed. Secondary outcomes will include the number of nominal days of breast pain (NDBP) 2 weeks before menstruation, WHOQOL-BREF scores, patient global assessment, breast glandular section thickness, and breast duct width three days before menstruation from baseline at weeks 12. This study will evaluate the effectiveness and safety of acupuncture to alleviate cyclic breast pain and to further explore the possible mechanisms underlying the effect.

DETAILED DESCRIPTION:
Sample size Sample size estimation was based on changes in the breast pain VAS(VAS-BP) score. According to the pre-trial, the VAS-BP score significantly decreased by 2.98 ±0.95 in MA group compared to 2.35 ±0.97 in the SM group after treatment from baseline. In the current trial, the investigators assume a significance level α = 0.05 and power (1-β) = 0.90, and providing for a two-sided outcome, at least 42 participants will be required for each group, as calculated by PASS version 11.0 (NCSS, LLC. Kaysville, UT, USA), assuming a two-tailed test with a 20% drop-out rate, a total of 108 patients (54 in each group) will be recruited.

Recruitment Patients are planned to be recruited via outpatient clinic, advertisements on websites and posters from hospitals and a chat group using WeChat (WeChat, Version: 8.0.21, Tencent, Shenzhen, China). Meanwhile, the investigators will cooperate with the gynecology and physical examination departments of the hospital for potential patients to ensure the target sample size is reached. All potentially eligible women with CM will be invited to the trial and be able to contact the researchers with the provided phone number. Patients who meet the inclusion criteria will be introduced to the study in detail and informed about the potential benefits and possible risks of this study, and will sign informed consent agreements.Then personal information including age, marriage, menstrual, and medical history and a series of questionnaire, ultrasound of breast, as recommended by SOGC guideline are cautiously recorded.

Data collection and management Plans for assessment and collection of outcomes The data will be collected using CRF. Questionnaires will be conducted by evaluators. The ultrasound image acquisition tests are performed by the ultrasound physicians. All data obtained during the study will be input into the database and anonymized and stored in the study folder. Only the research team has access to this particular research folder.

Plans to promote participant retention and complete follow-up The patients will receive sufficient information about the study and requirements during the recruitment. All patients will be reminded throughout the study to fill out the questionnaires during study visits.Throughout the follow-up period, the researchers will collect data and contact patients for completion. Patients are allowed to discontinue the study, the data collected up to the withdrawal date will be anonymized and used.

Data management The clinical trial management platform ResMan will be used to manage the data. Repeated input methods will be used to ensure that the entered data is correct. The database will be locked with a password, which will only be known by relevant personnel.

Statistical methods Statistical methods for primary and secondary outcomes The investigators will use SPSS 22.0 software(IBM SPSS Statistics; IBM Corp, Somers, NY)to perform all statistical analyses following the intention-to-treat principle. The CI will be established at 95%, and the significance level at 0.05. For continuous data, the data will be presented as mean±standard deviation when normally distributed or presented as median (IQR) when not normally distributed. Statistical comparisons will be performed by the independent-sample t tests or Wilcoxon rank-sum test for continuous data and by X2-test or Fisher exact test for categorical data, as appropriate. A p-value <0.05 will be considered statistically significant.

The investigators perform statistical analysis on complete case.The researcher will contact participants as much as possible to supplement missing data. The missing data will be assessed using an intention-to-treat analysis.

Oversight and monitoring In order to control the quality of the clinical trial, the study principal investigator and the coinvestigator will be responsible for the coordination, data management of each center monitoring.The study team will meet and discuss the problems in the the study every 3 months.Any decisions needing to be taken modifying the study will be done with the consensus of the entire study team after approval by the ethics committee of Pinggu Hospital of Beijing Traditional Chinese medicine hospital.

Adverse event reporting and harms All adverse events will be documented in the CRF throughout the trial. Adverse events related to acupuncture (such as severe pain, local hematoma, infection and abscess, and broken needles ), including discomfort after treatment, will be recorded in time and detail. A detailed description of the categories, severity and correlation with the treatment of the adverse events will be collected by patients themselves and evaluators. If the adverse event is severe and associated with the trial, the patient will be withdrawn from the study and given appropriate medical care.

Frequency and plans for auditing trial conduct The team will audit every 3 months. Pinggu Hospital of Beijing Traditional Chinese medicine hospital is the Trial Steering Committee and will supervise the trial. Beijing clinical research quality promotion center conducts an annual visit to check the existence and integrity of the investigation documents.

Plans for communicating important protocol amendments to relevant parties (e.g. trial participants, ethical committees) Any protocol amendments will be reported to the Ethics Committee of Pinggu Hospital of Beijing Traditional Chinese medicine hospital. Online trial registries will be updated accordingly.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-45 years old;
* Breast pain starts within 2 weeks before menses, and improves after onset, dull, heavy, or aching, bilateral, poorly localized, and extends into the axilla ;
* Fulfilling all conditions mentioned below: a. Moderate or severe breast pain as indicating 3 or more on scale of 1-10 on the VAS;b. History of CM for at least the past three consecutive cycles;c. Days of premenstrual breast pain≥3 days and≤14 days; d.A history of regular menstrual cycles of 28 plus/minus 3 days;
* Breast X-ray or breast ultrasound examination is excluded from malignant breast lesions;
* The patient signed the informed consent and voluntarily participated in the study.

Exclusion Criteria:

* Accepted acupuncture or drugs to treat breast pain within 1 month before entering the study;
* With breast inflammation, breast fibroma, breast cystic hyperplasia, and other benign breast lesions；
* With severe primary diseases in the cardiovascular system, pulmonary system, liver, kidney, and hematopoietic system;
* History of breast cancer among first-degree relatives;
* Breast pain caused by Costochondritis, chest wall injury, rib fracture, and other extramammary pain diseases;
* The patient is pregnant or lactating;
* with serious mental illness;
* Poor compliance;
* Patient has participated in other clinical trials within 1 month;
* with serious skin disease or infection at the acupuncture site.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 108 (Estimated)
Dates: Start 2022-07-20 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Breast Pain Visual Analog Scale score | from baseline at weeks 4, 8, 12,24,and36
  the change in the average ofBreast Pain Visual Analog Scale( VAS-BP )scores in the first 2 weeks of menstruation，The VAS-BP will be measured using a 10cm linear VAS with 0 representing no pain and 10 the worst imaginable pain, a higher score denotes more severe pain

SECONDARY OUTCOMES:
number of nominal days of breast pain | from baseline at weeks 4,8,12,24,and36
  The changes in the number of nominal days of breast pain (NDBP) during 2 weeks before menstruation
World Health Organization Quality Of Life Scale-Short Form | from baseline at weeks 12
  WHOQOL-BREF china version will be used to evaluate the QOL of the participants. The World Health Organization Quality Of Life Scale-Short Form( WHOQOL-BREF) Questionnaire consists of 26 items, in which the first and second questions of the questionnaire are about the QOL and health status in general. The next 24 questions assess the QOL in four dimensions: physical health (7items); psychological(6 items); environment (8 items); and social relationships (3 items). Each item is answered on a five-point scale. A higher score denotes a better quality of life.
breast glandular section thickness, and breast duct width | baseline at weeks 12
  Mammary ultrasonography will be used to observe breast glandular section thickness, and breast duct width three days before menstruation
Patients' global improvement assessment | at weeks 12
  It will be assessed by a 7-point self-reporting scale ranging from 1 to 7: significantly reduced, moderately reduced, slightly reduced, no change, slightly aggravated, moderately aggravated, and significantly aggravated. The proportion of patients reporting "significantly reduced" or "moderately reduced" is recorded as the response rate of overall efficacy

OTHER OUTCOMES:
Patients' acceptability toward acupuncture | at the end of the 1st treatment at week1 and the last treatment at week12.
  The acceptability of acupuncture will be assessed among participants in the MA group using a 3-point index: unacceptable (0 points), acceptable (1 point), and easy to accept (2 points). at the end of the week 1 and week12.
  ，
Blindness assessment | the last treatment session at week 12
  within 3 min after the last treatment session at week 12, all participants will be asked to answer the question do you think you have received acupuncture treatment and choose the answer between the options of Yes or No

CONTACTS AND LOCATIONS:
Overall Officials: Bin Shen, Study Director — Beijing Traditional Chinese Medicine Hospital Pinggu Hospital
Locations (1):
- Chuanyu, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
The data sharing will be available upon request and with permission and approval from the Pinggu Hospital of Beijing Traditional Chinese medicine hospital.
Supporting Information: CSR
Time Frame: After December 31, 2024

REFERENCES:
- [Derived] Yu C, Wang J, Shen B, Li X, Zhang R, Qin Y, Jian G, Guo J. Effectiveness of acupuncture in the treatment of cyclic mastalgia: a study protocol for a randomized controlled trial. BMC Complement Med Ther. 2022 Nov 18;22(1):297. doi: 10.1186/s12906-022-03779-8. PMID 36401325

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-05-28): https://cdn.clinicaltrials.gov/large-docs/77/NCT05408377/Prot_SAP_ICF_000.pdf